CLINICAL TRIAL: NCT01439503
Title: A Brief, Clinic-Based, Safer Sex Program for Young African-American Men
Brief Title: Safer Sex Program for Young African-American Men
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Richard Crosby (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor-Investigator, Richard Crosby, PhD/DDI Endowed Professor and Chair, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 11-0204-F3R; 1R01MH092226-01A1 (NIH)
Record Dates: First submitted 2011-09-20; First posted 2011-09-23 (Estimated); Last update posted 2019-02-21 (Actual); Status verified 2019-01

CONDITIONS: Gonorrhea; Chlamydia; Trichomoniasis; Syphilis; HIV Infections
MeSH Terms: conditions — Gonorrhea; Chlamydia Infections; Trichomonas Infections; Syphilis; HIV Infections | interventions — Methods

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Men receiving the control condition will be comprised of standard of care counseling from the clinic plus a variety of free condoms and water-based lubricants. They will also provide a specimen for STD testing, and receive text message questions for 12 weeks. The text messaging system will be used to collect self-reported dependent variables from men on a weekly basis. Texting will also serve as a constant method of contact between the PD and the enrolled men to remind them of follow-up assessments. In addition, the participants will complete the ACASI questionnaire to assess their sexual behavior, as well as demonstrate their condom application ability.
- Treatment (Experimental): Men receiving the treatment condition will receive text messages each week after their enrollment date and this will continue for 12 weeks to collect self-reported dependent variables. Text messaging will also be used to confirm and remind men about the day of each follow-up assessment. Each participant will also provide a specimen for STD testing, as well complete the ACASI questionnaire to assess sexual behavior and demonstrate their condom application ability. These participants will also be provided with a variety of free condoms and water-based lubricants. In addition, men in the treatment condition will also be enrolled in an education program.
  Interventions: Behavioral: Intervention

INTERVENTIONS:
Behavioral: Intervention — The intervention will consist of an education program. The education program includes providing the ability to enjoy condom use through improved skills related to finding the right "fit and feel" of condoms, using lubricants that are compatible with latex, negotiating condom use, negotiating sex, and talking with new and existing sex partners about ways to "sexualize" condoms.
  Arms: Treatment

SUMMARY:
To evaluate the efficacy of the adapted program a randomized controlled trial enrolling 620 eligible African American men who have sex with men (MSM) will be conducted. Men in the treatment condition will be compared to men receiving the control condition comprised of standard of care counseling from the clinic plus a free bag of condoms and water-based lubricants. This two-arm trial will test four hypotheses:

Aim: To test the efficacy of a brief, clinic-based and theory-guided, intervention designed to reduce STD incidence and risk of HIV acquisition/transmission among young African American men (15-29 years old) having sex with men and presenting for STD testing.

H1. Men randomized to receive the intervention will have a lower incidence rate of laboratory-confirmed STDs at each of three follow-up assessments compared to those receiving the control condition.

H2. Men randomized to receive the intervention will report significantly fewer acts of unprotected penetrative sex (penile-vaginal or penile-anal) between follow-up assessments compared to those receiving the control condition.

H3. Men randomized to receive the intervention will report having significantly fewer unprotected penetrative sex partners (for penile-vaginal or penile-anal sex) between follow-up assessments compared to those receiving the control condition.

H4. Men randomized to receive the intervention will report having significantly fewer negative experiences with condom use between follow-up assessments compared to those receiving the control condition.

H5. Men randomized to receive the intervention will demonstrate significantly greater improvement in condom application skills, throughout the 12-month study, compared to those receiving the control condition.

DETAILED DESCRIPTION:
The Centers for Disease Control and Prevention (CDC) has termed AIDS a "health crisis" for African Americans and has called for a heightened national response. The crisis is especially dramatic in the South and it is now apparent that young African American men who have sex with men (MSM) are exceedingly likely to be infected. Unfortunately, the ever-expanding HIV epidemic experienced by this population has not been matched by equal attention to the development of efficacious prevention programs. The proposed project expands upon an NIMH-funded study (R21 MH066682-01A1) conducted by Dr. Crosby. His study of young African American males found that a brief, clinic-based intervention reduced incidence of subsequent STDs by about 50%. This brief, one-on-one, intervention program, known as Focus on the Future (FOF), is a practical alternative to group-based safer sex programs that can be difficult to translate from science into practice. The program is now classified as a "Best Practice" intervention by CDC. This project will begin with an extensive formative phase designed to adapt FOF to MSM. The adapted program will seek to "sexualize" condoms to promote their consistent and correct use to better prevent STD/HIV. The program is uniquely flexible in that it can be applied to MSM regardless of their HIV serostatus. The adapted program will be tested by a two-arm efficacy trail. We will recruit 620 MSM (15-29 years of age) from a publicly-funded STD clinic in Jackson MS. Men in the treatment condition will be compared to men receiving the control condition comprised of standard of care counseling from the clinic plus a free ditty bag of supplies from the "condom and lube buffet" (condom/lube distribution). The trial will test four hypotheses: 1) Men randomized to receive the intervention will have a lower incidence rate of laboratory-confirmed STDs (by urine assay and rectal swab) at a 6-month and a 12-month follow-up assessment) compared to controls. 2) Men randomized to receive the intervention will report significantly fewer acts of unprotected penetrative sex (penile-vaginal or penile-anal) between follow-up assessments compared to controls. 3) Men randomized to receive the intervention will report having significantly fewer unprotected penetrative (penile-vaginal or penile-anal) sex partners between follow-up assessments compared to controls. 4) Men randomized to receive the intervention will report having significantly fewer negative experiences with condom use between follow-up assessments compared to controls. Given the dearth of evidence-based options for intervening with this vulnerable population in clinical settings, demonstrated efficacy of the adapted program has important implications for U.S. public health efforts directed towards the prevention of STD/HIV.

ELIGIBILITY:
Inclusion Criteria:

* 15-29 years of age
* Identifying as an African American Male
* Males must be presenting themselves for STD testing
* Males must report recently (past 3 months) engaging in penile-anal sex with other males as a "top" (meaning the insertive partner)

Exclusion Criteria:

* Males not identifying as African American
* Males older than 29 years of age
* Males that are not patients of the STD clinic
* Males who have not engaged in penile-anal sex with other males as a "top" within the past 3 months

Ages: 15 Years to 29 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 620 (Estimated)
Dates: Start 2012-09; Primary Completion 2017-11-25 (Actual); Study Completion 2018-04-02 (Actual)

PRIMARY OUTCOMES:
The frequency of unprotected sex rather than frequency of condom use will be used as the primary outcome measure. | 12 months (per participant)
  This will be achieved through the use of a centralized text messaging service. Once each week (throughout the 12-month observation period) men will receive questions, via text. The data from these weekly questions will be cumulated to form "3-month" variables that correspond with the STD-testing intervals between baseline and the first follow-up assessment and between the first follow-up assessment and the second one (at 6 months), as well as the "6-month" variables corresponding to the STD-testing interval between the 6-month assessment and the final assessment at 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Richard A Crosby, PhD, Principal Investigator — University of Kentucky; Leandro A Mena, MD, Principal Investigator — University of Mississippi Health Care
Locations (1):
- Mississippi State Department of Health STD Clinic, Jackson, Mississippi, United States